CLINICAL TRIAL: NCT02697708
Title: The Effect of Potatoes on Potassium Retention, Acid Base Balance, and Blood Pressure
Brief Title: Retention of Potassium From Potatoes and Potassium Gluconate, and the Effect on Blood Pressure.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Purdue University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1511016780
Record Dates: First submitted 2016-02-27; First posted 2016-03-03 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Hypertensive Disease
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will receive a controlled diet containing 2340 mg potassium.(K) During the 4 - 16 day phases they will receive an additional 0 mg K, 1000 mg K from potatoes, 1000 mg K from French Fries, and 1000 mg K from supplement in randomized order. Blood pressure will be measured every other day during the intervention. There will be a 2 week washout phase during each phase.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control Diet (Placebo Comparator): Control (no additional potassium added to diet): Arm will consist of a 16 day balance period with a basal diet set at ~2340mg K/day; based on average American intake.
  Interventions: Dietary Supplement: Potassium control diet
- Potassium Supplement Diet (Active Comparator): Potassium gluconate: Arm will consist of a 16 day balance period with the basal (control) diet plus the addition of 1000mg of K/day from potassium gluconate (12 tablets).
  Interventions: Dietary Supplement: Potassium gluconate diet
- Potato Diet (Experimental): Potato diet: Arm will consist of a 16 day balance period with a basal (control) diet with an addition of 1000mg of K/day from white potatoes.
  Interventions: Dietary Supplement: Potato Diet
- French fries Diet (Experimental): French fry diet: Arm will consist of a 16 day balance period with a basal (control) diet with an addition of 1000mg K/day from French fries.
  Interventions: Dietary Supplement: French Fries Diet

INTERVENTIONS:
Dietary Supplement: Potassium control diet — No additional potassium.
  Other Names: Control Diet
  Arms: Control Diet
Dietary Supplement: Potassium gluconate diet — 1000 mg K from potassium gluconate.
  Arms: Potassium Supplement Diet
Dietary Supplement: Potato Diet — 1000 mg K from potatoes.
  Arms: Potato Diet
Dietary Supplement: French Fries Diet — 1000 mg K from French Fries.
  Arms: French fries Diet

SUMMARY:
This study is designed to compare the effect of different dietary potassium sources on uptake and retention of potassium, as well as to determine the effect of potassium intake on blood pressure and acid-base balance. The study will compare three different sources of potassium given as a supplement, potatoes or French fries.

DETAILED DESCRIPTION:
Potassium is a shortfall nutrient according to the 2010 Dietary Guidelines for Americans. Only 3% of Americans meet the recommended Adequate Intake of 4700 mg/d for potassium. Average potassium intake is approximately half of the Recommended Dietary Allowance (RDA), with potatoes providing the highest percentage (19-20% of potassium) in the American diet. Recommended dietary potassium intakes were determined primarily to optimize protection against hypertension and secondarily to protect against stroke and coronary heart disease. In setting requirements for most minerals, bioavailability is usually considered. However, little is known about bioavailability of potassium and what is known is from supplements rather than food. Recently, we performed a potassium bioavailability study on white potatoes looking at 35 healthy, normotensive men and women at 3 levels of potassium intake as potatoes or potassium gluconate supplements. Bioavailability of potassium was determined from AUC of serial blood draws and cumulative urinary excretion. Serum potassium Area Under the Curve (AUC )increased with dose (P<0.0001) and did not differ due to source (p=0.52). Cumulative 24 h urinary potassium also increased with dose (p<0.0001) and was greater with potato than supplement (p<0.0001), concluding that bioavailability of potassium is as high from potatoes as from supplements. These data allow us to evaluate the quality of the food as a source of potassium. However, a remaining question is whether retention of potassium from potatoes is higher than from the salt, which requires a metabolic balance study to determine. The effects of potassium rich foods on blood pressure have also been recently accessed. A controlled feeding study would properly capture potassium retention and balance, as well as adequately control for any positive benefit potassium may have on blood pressure and other vascular outcomes.

Increasing potassium citrate decreased titratable acidity and improved calcium retention in a dose response manner in postmenopausal women. There is one Randomized Controlled Trial (RCT) of potassium on bone, in postmenopausal women, showing a benefit of a supplement of potassium chloride on protecting against bone loss. Similar studies have not been performed with food sources of potassium.

This study is designed to evaluate the effect of added potassium (K) from potatoes in the diet on K retention , blood pressure, and parameters related to bone health including calcium retention and acid base balance.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and above
* Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Pre-hypertensive, (SBP: 120-159mmHg).

Exclusion Criteria:

* Subjects taking more than one medication to treat hypertension
* Subject is taking medication to treat hypotension, or medication known to affect electrolyte metabolism or contain high levels of potassium or sodium, smoke cigarettes, use illegal drugs, or excessive alcohol intake.
* Current use systemic corticosteroids, androgens, phenytoin, erythromycin, thyroid hormones, lipid-lowering medication.
* Subjects who have hypertension (SBP > 160 mmHg), hypotension (SBP < 120mmHg) or diseases known to affect potassium metabolism (kidney disease or malabsorption disorders). History of myocardial infarction, diabetes mellitus, renal disease, gastrointestinal disease, pancreatitis, cholestatic liver disease, cancer.
* Subjects who are pregnant.
* Allergy or intolerance of intervention foods.
* Unwillingness to refrain from dietary supplements.
* Weight loss > 3kg in the past 2 months.
* Subjects with liver and/or lipid abnormalities (elevated alanine amino transferase (ALT) and aspartate amino transferase (AST), dyslipidemia).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 1, 3, 6, 8, 10, 12, 14, 16 days
  Systolic blood pressure measured directly three consecutive times after 15 min of supine rest.
Potassium balance/retention | Through out each day of each 16 day intervention
  Twenty four hour urine and feces will be collected on all intervention days of each phase. Urine will be analyzed for creatinine, K, Na, Ca, Mg according to the urine protocol. Some urine will be stored for future analysis and the rest discarded.
Potassium serum kinetics | Day 16 (24 hours) of each intervention period
  Following breakfast, which will include the respective source of potassium or control, pooled urine will be collected at 2, 4, 6, 12 and 24.h. Blood will be drawn (5ml each draw) at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6 and 24 hours post breakfast meal. , A catheter will be inserted in the arm at baseline and will be kept there until the blood draw at 6 hours. A needle will be used for the sample at 24 hours. BP will be measured after 4, 6, and 24h.

SECONDARY OUTCOMES:
Change in microcirculation | 1, and 16 days
  Vascular flow rate measured via Laser Doppler Flowmetry from right forearm for 60 min from the supine position.
Change in vascular flow rate | 1, 16 days
  Central blood pressure will be measured by pulse wave analysis. Measurements will be repeated at least three times within a 20 minute period after the subject has rested for at least 10 minutes in a seated position. The staff member will place a tonometer (pressure sensor) on the wrist to detect the radial pulse waveform. Measurements will be taken over the course of 5-15 minutes or until pulse wave signal reaches data acquisition parameters.
Acid-base balance | 14, 15 days
  Acid-base balance will be determined on two-end of phase 24 h urine collection to relate to urinary calcium and potassium excretion. Pre-prandial arterialized blood samples will be collected anaerobically using forearm venous blood from the heated hand (10) into a polypropylene syringe containing lyophilized lithium heparin. The blood samples will be stored at room temperature and analyzed within 1 h of collection. Renal acid-base balance will be measured using urinary Net Acid Excretion (NAE) and Potential Renal Acid Load (PRAL).

CONTACTS AND LOCATIONS:
Overall Officials: Connie Weaver, PhD, Principal Investigator — Purdue University, Nutrition Science
Locations (1):
- Department of Nutrition Science Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stone MS, Martin BR, Weaver CM. Short-Term Supplemental Dietary Potassium from Potato and Potassium Gluconate: Effect on Calcium Retention and Urinary pH in Pre-Hypertensive-to-Hypertensive Adults. Nutrients. 2021 Dec 9;13(12):4399. doi: 10.3390/nu13124399. PMID 34959951
- [Derived] Stone MS, Martin BR, Weaver CM. Short-Term RCT of Increased Dietary Potassium from Potato or Potassium Gluconate: Effect on Blood Pressure, Microcirculation, and Potassium and Sodium Retention in Pre-Hypertensive-to-Hypertensive Adults. Nutrients. 2021 May 11;13(5):1610. doi: 10.3390/nu13051610. PMID 34064968